CLINICAL TRIAL: NCT04851080
Title: Study of the Chronotype, Sleep Quality, Seasonal Pattern, Behavioral Time Preferences and the Functional State of the Body's Regulatory, Respiratory Systems in Individuals of Different Metabolic Status and Age
Brief Title: Medico-ecological Monitoring ((CSM, MCTQ, SPAQ, PSQI, HRV, Spirometry; Anthropometry, BP) of the Different Population Groups (Students, Schoolchildren, Volunteers) in North Caucasus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vladikavkaz Scientific Center of the Russian Academy of Sciences (Network)
Responsible Party: Sponsor
Other Study IDs: 1/7.20.03.21
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Conditionally Healthy Persons; Persons With a High Body Mass Index
Keywords: public health; metabolic syndrome; chronotype; sleep quality; seasonal pattern; regulatory systems; physiological stress
MeSH Terms: conditions — Metabolic Syndrome; Sleep Initiation and Maintenance Disorders | interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schoolchildren: Schoolchildren of Vladikavkaz secondary schools aged 13-16 years
  Interventions: Device: Heart Rate Variability; Device: Spirometry; Behavioral: Testing of psycho-physiological functions using four questionnaires
- Students: Students of North-Ossetian State Medical Academy at the age of 19-22 years
  Interventions: Device: Heart Rate Variability; Device: Spirometry; Behavioral: Testing of psycho-physiological functions using four questionnaires
- Volunteers: Scientists of the North Caucasian Research Institute of Mountain and Foothill Agriculture at the age of 30-56 years
  Interventions: Device: Heart Rate Variability; Device: Spirometry; Behavioral: Testing of psycho-physiological functions using four questionnaires

INTERVENTIONS:
Device: Heart Rate Variability — Heart rate variability is carried out using the complex of prenosological diagnostics "VARICARD 2.51" with the ISCIM 6.2 program is methodically based on the technology of analysis of heart rate variability, it uses the original scientific and theoretical substantiation of HRV indicators, which is based on modern ideas about stress, functional state of the body and assessment of health levels. It is designed to assess the risk of developing diseases in persons who are in states bordering health and disease. A decrease in the adaptive capabilities of the organism is considered as the main risk factor, the results obtained with its help are considered from the point of view of the level of health or stressful effects. It can be successfully used to control the effectiveness of medical intervention. Functionally, the complex is designed to register an electrical signal and form conclusions about the functional state of the body, assess the level of stress and its effect on health.
Device: Spirometry — Spirometry is carried out using the device Spirotest USPTs-01, equipped with liquid crystal indicators. It is non-invasive method for measuring air flows and volumes as a function of time using forced maneuvers. It is intended for functional diagnostics of the lungs, namely, indication and measurement of forced vital capacity and forced expiratory volume in the first second.
Behavioral: Testing of psycho-physiological functions using four questionnaires — Research of the behavioral time preferences by Composite Scale of Morningness (CSM, Smith C.S., Reilly C., Midkiff K., 1989). Translation into Russian by Kolomeichuk S., May 2015), of the chronotype by Munich ChronoType Questionnaire (MCTQ, Roenneberg T., Merrow M., LMU München, 2006, 2008. Translation into Russian by Putilov A.A., Danilenko K.V., approved by the authors October 2007, updated 2010), of the seasonal pattern by Seasonal Pattern Assessment Questionnaire (SPAQ, Rosenthal N.E., Genhart M., Sack D.A., Skwerer R.G., Wehr T.A., 1987.Translation into Russian by Putilov A.A., Danilenko K.V., Korneeva N.I. 1988, 2002), of the sleep quality by Pittsburgh Sleep Quality Index (PSQI, Russian edition Semenova E.A., Danilenko K.V., October 2009)

SUMMARY:
Observational Clinical Trial of the chronotype, sleep quality, seasonal pattern, behavioral time preferences, the functional state of the body's regulatory systems and respiratory systems in individuals of different age groups and metabolic status. In the process of medico-ecological monitoring, including all of the above, an assessment of the psycho-physiological status and the state of the regulatory and respiratory systems of the subjects' body, living in North Ossetia-Alania, will be made.

DETAILED DESCRIPTION:
Modern methods of medicine are aimed at maintaining homeostasis in a situation when, under the influence of factors of the external or internal environment, acute, chronical and extreme (in Covid-19 isolation) physiological stress, is formed, which the body is no longer able to compensate, and which forms the main group of human diseases - adaptation diseases, primarily cardiovascular, including cardiometabolic syndrome. Against the background of the Covid-19 pandemic, in conditions of limited physical activity, disruption of the daily routine and high psychophysiological load, various health disorders of both functional and organic nature may occur and existing pathologies may worsen.

The aim of the study - screening of health of different age categories of the population, based on research of chronotype, sleep quality, seasonal pattern, behavioral time preferences and functional state of body's regulatory and respiratory systems in individuals from the different age groups.

Methods: testing of psycho-physiological functions using Composite Scale of Morningness (CSM), Munich ChronoType Questionnaire (MCTQ), Seasonal Pattern Assessment Questionnaire (SPAQ), Pittsburgh Sleep Quality Index (PSQI); Heart rate variability (HRV); Spirometry; Anthropometry (measurement of height, weight, waist circumference), Blood pressure measurement (BP).

Statistical analyses planned to perform frequency, correlation, factorial and variance analyzes using Statistica 10,0 software ("StatSoft, Inc"). Data investigate by mean value (M) and standard deviation (SD) in case of normal data distribution or nonparametric method with determination of median (Me) and interquantile ranges (25th and 75th percentile) in the case of a distribution other than normal. ANOVA, MANOVA analysis. Statistically significant differences in all statistical tests set to P<0.05

ELIGIBILITY:
Inclusion Criteria:

conditionally healthy persons, persons with metabolic disorders in the presence of basic criterion MS - abdominal obesity.

Exclusion Criteria:

chronic somatic diseases; infectious diseases; malignant neoplasms of various organs and systems; viral infections; autoimmune diseases; mental illness; pregnancy and lactation in women

Ages: 13 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: population of the North Caucasus
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
H, (kg) | 5 minutes
  height
W, (m) | 5 minutes
  weight
WC (cm) | 5 minutes
  waist circumference
HR (beats per minute) - frequency of the pulse | 5 minutes
  average pulse rate over the observation period, which integrally characterizes the level of functioning of the circulatory system.
SDNN, (ms) - standard deviation of all NN intervals | 5 minutes
  reflects all the cyclic components responsible for variability and the total effect of autonomic regulation of blood circulation
RMSSD, (ms) - square root of the mean of the sum of the squares of differences between adjacent NN intervals | 5 minutes
  measurements of short-term variation, estimate high frequency variations in heart rate and activity of the parasympathetic link of regulation.
pNN50, (ms) | 5 minutes
  the proportion derived by dividing NN50 by the total number of NN intervals, where NN50 - number of pairs of adjacent NN intervals differing by more than 50 ms in the entire recording
LF, (ms2) - power in low frequency range (0.04-0.15 Hz) | 5 minutes
  reflects the state of the sympathetic from the case of the ANS, and, in part, the parasympathetic department
HF, (ms2) - power in high frequency range (0.15-0.4 Hz) | 5 minutes
  reflects the parasympathetic link of regulation
LF/HF - ratio LF (ms2)/HF (ms2) | 5 minutes
  reflects the ratio of the levels of activity of the central and autonomous circuits of regulation
TP, (ms2) - total power of the heart rate variability spectrum | 5 minutes
  reflects the total power of the heart rate variability spectrum
FVCL, (liter) - forced vital capacity of lungs | individually (at least six seconds)
  qualifies the maximum volume of air that a person can exhale after taking the deepest possible breath
FEV1, (liters per second) - forced expiratory volume in the first second of the forced expiratory maneuver | 1 second
  is an indicator of the mechanical properties of the ventilation apparatus, reflecting the total patency of the airways, elastic properties of the lungs and chest
mun-wd-fas (hours:minutes) - falling asleep time on working days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-wd (hours:minutes) - sleep duration on working days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-wd-mid (hours:minutes) - middle of sleep duration on working days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-wd-wut (hours:minutes) - wake up time on working days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-fd-fas (hours:minutes) - falling asleep time on weekend days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-fd (hours:minutes) - sleep duration on weekend days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-fd-mid (hours:minutes) - middle of sleep duration on weekend days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
mun-fd-wut (hours:minutes) - wake up time on weekend days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
DEW (hours:minutes) - daylight exposure on working days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
DEF (hours:minutes) - daylight exposure on weekend days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
JLW (hours:minutes) - jet lag on working days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
JLF (hours:minutes) - jet lag on weekend days | about 10-15 minutes on each Questionnaire
  Parameters of Munich ChronoType Questionnaire (MCQT) (primary outcome measures 15-25) documenting individual sleep time, self-assessment of illumination and self-assessment of chronotype, taking into account work and days off separately. Sleep time is a good indicator for chronotype when adjusted for the amount of sleep received during the workweek and on weekends, as well as the amount of time subjects spend outdoors in daylight.
C1 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Daytime mood": how much (score) of a problem has it been to keep up enthusiasm to get things done during the past month
C2 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Sleep latency": minutes to fall asleep each night (≤15min=0; 16-30 min=1; 31-60 min=2, >60 min=3) + how often a person cannot fall asleep within 30 minutes (if sum is equal 0=0; 1-2=1; 3-4=2; 5-6=3)
C3 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Sleep duration": hours of actual sleep at night (>7=0; 6-7=1; 5-6=2; <5=3)
C4 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Sleep efficiency": (total of hours asleep)/(total of hours in bed) x 100; >85%=0, 75%-84%=1, 65%-74%=2, <65%=3
C5 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Sleep disturbance": sum of Component 5b-5j scores (0=0; 1-9=1; 10-18=2; 19-27=3)
C6 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Subjective sleep quality": self-reported sleep quality over the past month
C7(score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  "Sleeping pills and daytime sleepiness": how often a person take medicine to help asleep during the past month+ how often a person had trouble staying awake while driving, eating meals, or engaging in social activity during the past month
Global PSQI Score = C1+C2+C3+C4+C5+C6+C7 | about 10-15 minutes on each Questionnaire
  Each component is scored from 0 to 3 points, forming an overall PSQI score ranging from 0 to 21, where higher scores indicate poorer sleep quality. PSQI is useful for determining good and bad sleep quality. An overall PSQI score above 5 indicates poor sleep.
CMQ (score) - Component of Composite Scale of Morningness | about 10-15 minutes on each Questionnaire
  Composite Scale of Morningness characterize in the form of questions: morning activity, morning affects and eveningness. CSM ask mostly for preferred time of day and imply answers based on clock times or comparisons with others in a given population. In CSM regarding preferred sleeping and waking times, respondents select the most suitable option from a list of time increments. Issues like ease of waking, alertness throughout the day, and exercise are also queried. Potential scores for the scale's items range from 1 to 4 or 5, with higher scores indicating a greater degree of morningness. Cutoffs for the scale were chosen using the upper and lower percentiles of the scale: A score of 22 or below indicates an evening type, a score above 44 indicates a morning type, and scores in between receive a classification of intermediate. In total we used two parameters: CMQ - sum of the scores of the scale's items range; CSMN - nominal chronotype rating.
CSMN (nominal) - Component of Composite Scale of Morningness | about 10-15 minutes on each Questionnaire
  Composite Scale of Morningness characterize in the form of questions: morning activity, morning affects and eveningness. CSM ask mostly for preferred time of day and imply answers based on clock times or comparisons with others in a given population. In CSM regarding preferred sleeping and waking times, respondents select the most suitable option from a list of time increments. Issues like ease of waking, alertness throughout the day, and exercise are also queried. Potential scores for the scale's items range from 1 to 4 or 5, with higher scores indicating a greater degree of morningness. Cutoffs for the scale were chosen using the upper and lower percentiles of the scale: A score of 22 or below indicates an evening type, a score above 44 indicates a morning type, and scores in between receive a classification of intermediate. In total we used two parameters: CMQ - sum of the scores of the scale's items range; CSMN - nominal chronotype rating.
SSI (score) - Component of Seasonal Pattern Assessment Questionnaire | about 10-15 minutes on each Questionnaire
  seasonality index (sum of test score of Component 11 of Seasonal Pattern Assessment Questionnaire)
SAD (nominal) - Component of Seasonal Pattern Assessment Questionnaire - seasonal affective disorder | about 10-15 minutes on each Questionnaire
  nominal finding of the seasonal affective disorder
selfSAD (nominal) - Component of Seasonal Pattern Assessment Questionnaire | about 10-15 minutes on each Questionnaire
  self-assessment by the subject of changes in his state depending on the season

SECONDARY OUTCOMES:
SI (c.u.)- stress index, | 5 minutes
  reflects the degree of stress in regulatory systems.
IC (c.u.)- centralization index, | 5 minutes
  reflects the degree of activity of central regulation circuit
PHF, (%) - power of the spectrum of the high-frequency component of variability in % of the total power of oscillations | 5 minutes
  evaluates the relative level of activity of the parasympathetic link of regulation
PLF, (%) - power of the spectrum of the low-frequency component of variability in% of the total power of oscillations | 5 minutes
  evaluates the relative level of activity of the vasomotor center
PVLF, (%) - power of the spectrum of the very low-frequency component of variability in% of the total power of oscillations | 5 minutes
  evaluates the relative level of activity of the sympathetic link of regulation
psqi10 (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  having a roommate
psqi11 (a-e) (score) - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  ask your roommate how often you have: (a)loud snoring, (b) prolonged breath holding during sleep, (c) episodes of disorientation during sleep, (d) other manifestations of anxiety during sleep
psqi11cause - Component of Pittsburgh Sleep Quality Index | about 10-15 minutes on each Questionnaire
  describe other manifestations of anxiety during sleep

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Sergeevna Datieva, MD, Principal Investigator — Vladikavkaz Scientific Centre of the Russian Academy of Sciences
Locations (1):
- Institute of Biomedical Investigations - the Affilliate of Vladikavkaz Scientific Centre of the Russian Academy of Sciences, Vladikavkaz, RNO-Alania, Russia

IPD SHARING:
Plan to Share IPD: No